CLINICAL TRIAL: NCT02124460
Title: Improving Childhood Obesity Outcomes: Testing Best Practices of Positive Outliers
Brief Title: Connect 4 Health: An Intervention to Improve Childhood Obesity Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Vanguard Medical Associates (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Academic Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IH-1304-6739
Record Dates: First submitted 2014-04-14; First posted 2014-04-28 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-02

CONDITIONS: Overweight; Obesity
Keywords: Pediatric; Obesity; Overweight; Intervention
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Primary Care (No Intervention): We will provide current "best practice" to the control arm. Patients with a BMI greater than or equal to the 85th percentile will be flagged in the electronic health record. Clinicians are also provided with clinical decision support tools for pediatric weight management. We will encourage providers to schedule a follow up visit for weight management or make a referral to Harvard Vanguard Medical Associates nutritionists for children in this arm. We will also provide this group with a community resource guide and educational text messages.
- Health Coaching (Experimental): The intervention for this study will consist of the same best practices received by the enhanced primary care group well as the following three elements: visits with a health coach, connection to community resources and an interactive text messaging program.
  Interventions: Behavioral: Health Coaching

INTERVENTIONS:
Behavioral: Health Coaching — Parent/child duos enrolled in the intervention group will participate in a total of six visits with a trained health coach. During these visits, the health coach will coach the parent/child duos on improving obesity-related behaviors .
  The health coach will also help the family identify supports to assist with behavior change; discuss family health habits and the home environment; and review and encourage use of materials related to both specific target behaviors and available resources in the community.
  Following the first call with the health coach, parents will receive semi-weekly text messages designed by the study team. The messages will alternate in structure between 2 types of messages; 1) skills training messages will deliver tips and motivational messages to help their child practice the study's goals and 2) self monitoring messages will ask parents to respond to the message and track health behaviors important to this study.
  Arms: Health Coaching

SUMMARY:
Health care system (HCS)-based interventions have been limited by their inattention to social and environmental barriers that impede improvement in obesity-related behaviors. Additionally, current pediatric obesity care delivery relies on an outdated provider:patient paradigm which is ill-suited for a problem as prevalent as obesity. HCSs often lack the organizational structure to provide longitudinal care for children with chronic illnesses, the clinicians to manage and support patients with chronic illnesses outside of clinic, and/or the health information systems that support the use of evidence-based practices at the point-of-care. Thus, the research question this study is designed to address is whether a novel approach to care delivery that leverages delivery system and community resources and addresses socio-contextual factors will improve family-centered childhood obesity outcomes.

The primary specific aims are to examine the extent to which the intervention, compared to the control condition, results in:

1. A smaller age-associated increase in BMI over a 12-month period.
2. Improved parental and child ratings of pediatric health-related quality of life.

The secondary aims are:

1. To examine parental ratings of quality and family-centeredness of pediatric obesity care and compare outcomes among participants in the intervention with the control condition
2. To assess change in weight-related behaviors and compare outcomes among participants in the intervention with the control condition
3. To assess the following process measures:

   * Reach
   * Extent of implementation
   * Fidelity to protocol
   * Parent satisfaction
4. To examine the extent to which neighborhood environments modify observed intervention effects
5. To assess the documentation of Healthcare Effectiveness Data and Information Set (HEDIS) measures in participant medical records

ELIGIBILITY:
Inclusion Criteria:

* child is age 2.0 through 12.9 years at baseline primary care visit,
* child's BMI is equal to or exceeds the 85th percentile for age and sex at baseline primary care visit,
* at least 1 parent has an active email address,
* at least one parent is comfortable reading and speaking in English.

Exclusion Criteria:

* children who do not have at least one parent/legal guardian who is able to follow study procedures for 1 year,
* families who plan to leave HVMA within the study time frame,
* families for whom the primary care clinician thinks the intervention is inappropriate, e.g., emotional or cognitive difficulties,
* children who have a sibling already enrolled in the study,
* children with chronic conditions that substantially interfere with growth or physical activity participation.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 721 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsie M Taveras, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Harvard Vanguard Medical Associates, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Simione M, Ferreira P, Luo M, Hoover C, Perkins M, Fiechtner L, Taveras EM. Psychometrics of the modified family-centered care assessment short version for childhood obesity. Health Qual Life Outcomes. 2024 Sep 2;22(1):71. doi: 10.1186/s12955-024-02284-5. PMID 39218948
- [Derived] Simione M, Ferreira P, Luo M, Hoover C, Perkins M, Fiechtner L, Taveras EM. Psychometrics of the modified Family-Centered Care Assessment short version for childhood obesity. Res Sq [Preprint]. 2024 May 15:rs.3.rs-4365570. doi: 10.21203/rs.3.rs-4365570/v1. PMID 38798356
- [Derived] Simione M, Sharifi M, Gerber MW, Marshall R, Avalon E, Fiechtner L, Horan C, Orav EJ, Skelton J, Taveras EM. Family-centeredness of childhood obesity interventions: psychometrics & outcomes of the family-centered care assessment tool. Health Qual Life Outcomes. 2020 Jun 11;18(1):179. doi: 10.1186/s12955-020-01431-y. PMID 32527270
- [Derived] Baskind MJ, Taveras EM, Gerber MW, Fiechtner L, Horan C, Sharifi M. Parent-Perceived Stress and Its Association With Children's Weight and Obesity-Related Behaviors. Prev Chronic Dis. 2019 Mar 28;16:E39. doi: 10.5888/pcd16.180368. PMID 30925139
- [Derived] Bala N, Price SN, Horan CM, Gerber MW, Taveras EM. Use of Telehealth to Enhance Care in a Family-Centered Childhood Obesity Intervention. Clin Pediatr (Phila). 2019 Jun;58(7):789-797. doi: 10.1177/0009922819837371. Epub 2019 Mar 20. PMID 30894004
- [Derived] Fiechtner L, Puente GC, Sharifi M, Block JP, Price S, Marshall R, Blossom J, Gerber MW, Taveras EM. A Community Resource Map to Support Clinical-Community Linkages in a Randomized Controlled Trial of Childhood Obesity, Eastern Massachusetts, 2014-2016. Prev Chronic Dis. 2017 Jul 6;14:E53. doi: 10.5888/pcd14.160577. PMID 28682745
- [Derived] Taveras EM, Marshall R, Sharifi M, Avalon E, Fiechtner L, Horan C, Gerber MW, Orav EJ, Price SN, Sequist T, Slater D. Comparative Effectiveness of Clinical-Community Childhood Obesity Interventions: A Randomized Clinical Trial. JAMA Pediatr. 2017 Aug 7;171(8):e171325. doi: 10.1001/jamapediatrics.2017.1325. Epub 2017 Aug 7. PMID 28586856
- [Derived] Taveras EM, Marshall R, Sharifi M, Avalon E, Fiechtner L, Horan C, Orav J, Price SN, Sequist T, Slater D. Connect for Health: Design of a clinical-community childhood obesity intervention testing best practices of positive outliers. Contemp Clin Trials. 2015 Nov;45(Pt B):287-295. doi: 10.1016/j.cct.2015.09.022. Epub 2015 Sep 30. PMID 26427562

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Primary Care: We will provide current "best practice" to the enhanced primary care arm. We will encourage providers use clinical decision support tools and to schedule a follow up visit for weight management or make a referral to Harvard Vanguard Medical Associates nutritionists for children in this arm. We will also provide this group with a community resource guide and educational text messages.
- Health Coaching: The intervention group will receive the same components as the enhanced primary care group for this study plus the following elements: visits with a health coach, individualized connection to community resources and an interactive text messaging program.
  Parent/child duos enrolled in the intervention group will participate in a total of six visits with a trained health coach. The health coach will coach the parent/child duos on improving obesity-related behaviors and help the family identify supports to assist with behavior change and encourage use of materials related to both specific target behaviors and available resources in the community.
  Parents will receive semi-weekly text messages. The messages will alternate in structure between 1) skills training messages will deliver tips to help their child practice the study's goals and 2) self monitoring messages will ask parents to respond and track health behaviors important to this study.
Period: Overall Study
Arm/Group | Enhanced Primary Care | Health Coaching
Started | 361 | 360
Completed | 328 | 336
Not Completed | 33 | 24

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Primary Care: Arm: No Intervention: Enhanced Primary Care We will provide current "best practice" to the control arm. We will encourage providers to schedule a follow up visit for weight management or make a referral to Harvard Vanguard Medical Associates nutritionists for children in this arm. We will also provide this group with a community resource guide and educational text messages.
- Health Coaching: Arm: Experimental: Health Coaching The intervention for this study will consist of three elements: visits with a health coach, connection to community resources and an interactive text messaging program.
- Total: Total of all reporting groups
Arm/Group | Enhanced Primary Care | Health Coaching | Total
Number analyzed (Participants) | 361 | 360 | 721
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 361 | 360 | 721
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.0 (3.0) | 8.1 (3.0) | 8.0 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 180 | 368
  Male | 173 | 180 | 353
Region of Enrollment [Number; unit: participants]
  United States | 361 | 360 | 721
BMI z score [Mean (Standard Deviation); unit: BMI z score units] | 1.90 (0.51) | 1.86 (0.52) | 1.88 (0.52)
Pediatric Quality of Life (PedsQL) Summary Score [Mean (Standard Deviation); unit: units on a scale] — Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better HRQOL. Scale Scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). If more than 50% of the items in the scale are missing, the Scale Score is not computed.
  units on a scale | 86.0 (10.8) | 85.4 (11.4) | 85.7 (11.1)
Parent Resource Empowerment [Mean (Standard Deviation); unit: units on a scale] — The five items in the scale assessed parents' perceived knowledge of resources, ability to access resources, comfort with accessing resources, knowledge of how to find resources, and ability to acquire resources related to child weight management. Responses ranged from Strongly disagree to Strongly agree (range = 1-4). Items were averaged to create a summary parental resource empowerment score (range= 1-4), where a higher score indicated greater perceived knowledge and ability to access resources related to weight management. Cronbach's α for this score was 0.87.
  units on a scale | 2.93 (0.59) | 2.96 (0.53) | 2.95 (0.56)

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI z Score
Description: Height and weight will be measured by the medical assistants at each site using standard protocols. BMI measures will be obtained from the electronic health record (EHR) as provided through usual care. BMI measures will be converted to z-scores using CDC age and sex-specific normative data for children between 2 and 20 years old. This will allow the research team to combine data across children of different ages.
Time Frame: baseline and one year
Measure: Mean (95% Confidence Interval); unit: BMI z score units
Groups:
- Enhanced Primary Care: We will provide current "best practice" to the control arm. Patients with a BMI greater than or equal to the 85th percentile will be flagged by in the electronic health record. Clinicians are also provided with clinical decision support tools for pediatric weight management. We will encourage providers to schedule a follow up visit for weight management or make a referral to Harvard Vanguard Medical Associates nutritionists for children in this arm. We will also provide this group with a community resource guide and educational text messages.
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
BMI z score units | -0.06 [-0.10 to -0.02] | -0.09 [-0.13 to -0.05]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = 0.3928, Linear repeated measures; Multiple imputation was used for missing follow-up data; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.08 to 0.03] — Health Coaching group compared to Enhanced Primary Care

2. Primary Outcome: Change in Quality of Life
Description: The PedsQL is an extensively validated, widely used, 23-item measure of health-related quality of life in children with chronic conditions such as obesity. Parents will be asked to complete 4 subscales: physical health, school, social, and emotional functioning which exists for parental report of children as young as 2 years of age. Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), so that higher scores indicate better HRQOL. Scale Scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). If more than 50% of the items in the scale are missing, the Scale Score is not computed.
Time Frame: baseline and one year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
units on a scale | 0.65 [-0.38 to 1.67] | 1.53 [0.51 to 2.56]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = 0.2306, Linear repeated measures; Multiple imputation used for missing data at follow-up; Mean Difference (Net) = 0.89, 95% CI 2-sided [-0.56 to 2.33] — Health Coaching group compared to Enhanced Primary Care

3. Primary Outcome: Change in Parent Resource Empowerment
Description: The five items in the scale assessed parents' perceived knowledge of resources, ability to access resources, comfort with accessing resources, knowledge of how to find resources, and ability to acquire resources related to child weight management. For each question, parents responded strongly disagree, disagree, agree, or strongly agree, which were worth 1 to 4 points, respectively. Items were averaged to create a summary parental resource empowerment score (range= 1-4), where a higher score indicated greater perceived knowledge and ability to access resources related to weight management. Cronbach's α for this score was 0.87.
Time Frame: Baseline to one-year follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
units on a scale | 0.29 [0.22 to 0.35] | 0.22 [0.15 to 0.29]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = .14, Linear repeated measures; Multiple imputation used for missing data at follow-up; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.02 to 0.16] — Health Coaching group compared to Enhanced Primary Care

4. Secondary Outcome: Change in Screen Time
Description: Average hours/day spent watching television, videos, or playing games displayed on media such as television, desktop computers, laptops, portable DVD players, iPads or smartphones.
Time Frame: baseline and one year
Measure: Mean (95% Confidence Interval); unit: hours/day
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
hours/day | -0.06 [-0.12 to 0.00] | -0.56 [-0.78 to -0.34]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = 0.0016, Linear repeated measures; Multiple imputation used for missing data at follow-up; Mean Difference (Net) = -0.50, 95% CI 2-sided [-0.81 to -0.19]

5. Secondary Outcome: Change in Sleep
Description: Average hours/day spent sleeping
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: hours/day
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
hours/day | -0.02 [-0.16 to 0.12] | 0.40 [0.25 to 0.55]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p < .0001, Linear repeated measures — Multiple imputation used for missing data at follow-up; Mean Difference (Net) = 0.42, 95% CI 2-sided [0.22 to 0.62]

6. Secondary Outcome: Change in Physical Activity
Description: In the past week, how many days the child was physically active for a total of at least 60 minutes per day.
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: days/week
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
days/week | 0.15 [-0.10 to 0.40] | 0.33 [0.09 to 0.58]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = 0.3043, Linear repeated measures; Multiple imputation used for missing data at follow-up; Mean Difference (Net) = 0.18, 95% CI 2-sided [-0.16 to 0.53]

7. Secondary Outcome: Change in Fruit and Vegetable Consumption
Description: Number of times the child consumed of vegetables and fruits yesterday
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: times/day
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
times/day | 0.19 [0.01 to 0.36] | 0.50 [0.33 to 0.68]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = 0.0113, Linear repeated measures; Multiple imputation used for missing data at follow-up; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [0.07 to 0.56]

8. Secondary Outcome: Change in Consumption of Sugar-sweetened Beverages and Juice
Description: Number of time child consumed juice (e.g., orange juice, apple juice, or grape juice), fruit-flavored drinks (e.g., Kool-Aid, sports drinks, Goya juice, etc.), regular soda, soft drinks, or Malta yesterday.
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: times/day
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 361 | 360
times/day | -0.03 [-0.20 to 0.14] | -0.25 [-0.41 to -0.08]
Statistical Analysis 1: Comparison: Enhanced Primary Care vs Health Coaching; Test type: Superiority or Other; p = 0.0792, Linear repeated measures; Multiple imputation used for missing data at follow-up; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.45 to 0.03]

9. Post Hoc Outcome: Increased Satisfaction With Care at Harvard Vanguard Medical Associates (HVMA)
Description: This is a feasibility and acceptability measure from the study.
Time Frame: 1 year
Population: The number of participant analyzed was based only on those who completed the follow-up survey (as the questions were not asked at baseline) and excluded those with missing responses.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 321 | 315
Participants | 153 | 199

10. Post Hoc Outcome: Parent Very Satisfied With Content of Connect 4 Health Text Messages or Emails.
Description: This is a feasibility and acceptability measure from the study.
Time Frame: 1 year
Population: The number of participant analyzed was based only on those who completed the follow-up survey (as the questions were not asked at baseline) and excluded those with missing responses. Additionally, only those who responded Yes to the previous question asking if they received text messages were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 292 | 313
Participants | 156 | 226

11. Post Hoc Outcome: Received Information From Connect 4 Health About Resources in the Community
Description: This is a feasibility and acceptability measure from the study.
Time Frame: 1 year
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 323 | 315
Participants | 195 | 301

12. Post Hoc Outcome: Received Text Messages or Emails From Connect 4 Health
Description: This is a feasibility and acceptability measure from the study.
Time Frame: 1 year
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 323 | 315
Participants | 295 | 314

13. Post Hoc Outcome: Parent Very Satisfied With Information he/She Received About Resources in the Community
Description: This is a feasibility and acceptability measure from the study.
Time Frame: 1 year
Population: The number of participant analyzed was based only on those who completed the follow-up survey (as the questions were not asked at baseline) and excluded those with missing responses. Additionally, only those who responded Yes to the previous question asking if they received community resources were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Primary Care | Health Coaching
Number analyzed (Participants) | 195 | 301
Participants | 128 | 228

ADVERSE EVENTS:
Arm/Group | Enhanced Primary Care | Health Coaching
Serious Adverse Events (participants affected / at risk) | 0/361 | 0/360
Other Adverse Events (participants affected / at risk) | 0/361 | 0/360

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No